CLINICAL TRIAL: NCT05240235
Title: The Effect of Manual Lymph Drainage in the Treatment of Breast Edema That May Occur in Patients Undergoing Breast-conserving Surgery and Adjuvant Radiotherapy-Randomized Controlled Study
Brief Title: The Effect of Manual Lymph Drainage in the Treatment of Breast Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATADEK-2023/18
Record Dates: First submitted 2022-01-26; First posted 2022-02-15 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer and Rehabilitation
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education, compression and exercise therapy (Active Comparator): Patients will be given exercise therapy every day for the first two weeks. Afterwards, patients will be taken to the same therapy in the hospital for 1 day a week, and on other days they will do home exercise at home for 10 minutes.
  Interventions: Other: Education, compression and exercise therapy
- Education, compression,exercise therapy and manual lymph drainage (Active Comparator): Patients will be given manual lymph drainage for one and a half hours every day for the first two weeks. Afterwards, patients will be taken to the same therapy in the hospital for 1 day a week, and on other days they will do self manual lymph drainage at home for 10 minutes.
  Interventions: Other: Education, compression and exercise therapy manual lymph drainage

INTERVENTIONS:
Other: Education, compression and exercise therapy — Education; It includes information about the disease, information about risk factors, information that one should pay attention to, and skin care. For compression, sponge-shaped pads that create compression into the bra and prepared by the lymphedema physiotherapist will be used. The exercises will include breathing and upper extremity joint movement exercises determined by Casley-Smith, and the other days to be applied by the physiotherapist when the patient comes to the session will be applied by the patient once a day at home.
  Arms: Education, compression and exercise therapy
Other: Education, compression and exercise therapy manual lymph drainage — Education; It includes information about the disease, information about risk factors, information that one should pay attention to, and skin care. For compression, sponge-shaped pads that create compression into the bra and prepared by the lymphedema physiotherapist will be used. The exercises will include breathing and upper extremity joint movement exercises determined by Casley-Smith, and the other days to be applied by the physiotherapist when the patient comes to the session will be applied by the patient once a day at home. In addition, patients will be given manual lymph drainage for one and a half hours every day for the first two weeks. Afterwards, patients will be taken to the same therapy in the hospital for 1 day a week, and on other days they will do self manual lymph drainage at home for 10 minutes.
  Arms: Education, compression,exercise therapy and manual lymph drainage

SUMMARY:
Breast conserving surgery (BCS) is widely used in the treatment of breast cancer. Breast edema can be seen frequently after BCS and radiotherapy applications. Breast edema affects quality of life and may result in a cosmetically unsatisfactory outcome for the patient. Therefore, it is important to treat and prevent its development. In the light of this information, the present randomized controlled study aims to determine the effect of manual lymph drainage method in the treatment of breast edema in patients undergoing breast-conserving surgery and adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent breast-conserving surgery and received adjuvant radiotherapy
2. Patients with Sentinel Lymph Node Biopsy or axillary lymph node dissection
3. Female patients between the ages of 18-75
4. Patients who cannot read and write Turkish

Exclusion Criteria:

1. A previous cancer
2. Decompensated heart failure
3. Untreated congestive heart failure
4. Active infection
5. Uncontrolled hypertension
6. Acute kidney failure
7. Patients with acute deep vein thrombosis
8. Metastasis and/or recurrence during treatment
9. Patients who have undergone another surgery related to the breast and chest area
10. Patients who develop lymphedema in the upper extremity during therapy will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
LENT-SOMA criteria in breast edema | Change from baseline LENT-SOMA criteria at 12 weeks
  Breast Cancer Conservative treatment core objective measurement. It has a score between 13-52 points. As the score increases, it is seen that breast edema worsens. A decrease in the score indicates improvement in breast edema.
Breast edema questionnaire | Change from baseline breast edema questionnaire at 12 weeks
  Getting 8.5 points from the questionnaire is the cut-off point. There is no breast edema below 8.5, there is breast edema above 8.5. It has a score between 0-80 points.
Clinical features of breast cancer and breast edema | Change from baseline clinical features of breast cancer and breast edema at 12 weeks
  The presence of breast fibrosis or edema, teleangiectasia or dyspigmentation will be scored on a 4-point categorical scale. The scale will be in the range of 0-16 points, high scores will indicate worsening of breast edema, and low scores will indicate improvement.
Qualitiy of Life - European Organization for Research and Treatment of Cancer EORTC- BR23 | Change from baseline Quality of life (EORTC- BR23) test at 12 weeks
  The EORTC-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.All scores will linearly transforme to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score. More severe symptoms or problems are represented by high symptom scores or items.

SECONDARY OUTCOMES:
Breast pain intensity will be measured with the Visual Analog Scale | Change from baseline Visual Analog Scale test at 12 weeks
  The scale is 10 cm long and is applied by specifying a point on the vertical or horizontal line with two different ends (0 = no pain, 10 = the most severe pain) corresponding to the severity of pain felt by the patient.
Quality of life test (EORTC QOL-C30) | Change from baseline Quality of life test (EORTC QOL-C30) at 12 weeks
  It includes 30 items that are grouped into five scales functional (physical, social, emotional functioning, cognitive and role), three scales of symptoms (fatigue, pain, nausea and vomiting), a global scale of health / quality of life and a number of related individual items with the symptoms of the disease and its treatment, as well as an item of economic impact. The answers to the items on the scales refer to "last week," except the patient's physical functioning scale whose time frame is the present. These answers they obey a Likert format, which ranges from 1 ("Not at all") and 4 ("A lot")

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided